CLINICAL TRIAL: NCT01369758
Title: MyoSure Hysteroscopic Tissue Removal System Registry Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMP 200905
Record Dates: First submitted 2010-11-11; First posted 2011-06-09 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Uterine Fibroids; Polyps
Keywords: morcellator; hysteroscope; myomectomy; polypectomy; uterine fibroids; uterine polyps
MeSH Terms: conditions — Leiomyoma; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intrauterine pathology, myomectomy (Experimental): Subjects with intrauterine fibroids and/or polyps will undergo intrauterine pathology removal using the MyoSure Tissue Removal System; myomectomy procedure.
  Interventions: Device: MyoSure Tissue Removal System

INTERVENTIONS:
Device: MyoSure Tissue Removal System — The MyoSure Tissue Removal Device consists of a hand-held tissue removal device comprising a mechanical drive assembly connected to a drive cable and associated control box on one end, and a 3 mm shaft on the other end of the device. The shaft is approximately 12 cm long and equipped with an open channel that houses an oscillating blade. When the side channel is exposed to target tissue and the motor is activated, the oscillating blade will cut the tissue within the channel. Once cut, the tissue travels down the center of the 3mm shaft via suction coupled to the proximal end of the tissue removal device, and is trapped in a vacutainer bottle.
  Other Names: Myomectomy procedure

SUMMARY:
The objective of this study is to demonstrate the safety and effectiveness of community gynecologist initiated treatment of intra-uterine polyps and submucosal fibroids with the MyoSure Hysteroscopic Tissue Removal System in a significantly sized patient population.

DETAILED DESCRIPTION:
Between 500 and 600 subjects will be enrolled in a prospective, multi-center registry study. Approximately 100 of these cases will be completed in an office setting, with the remaining 400-500 cases completed in a hospital outpatient or ambulatory surgery center. Subjects will undergo a hysteroscopic tissue removal procedure to remove intrauterine polyps and submucosal fibroids.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female between 18 and 65 years of age
2. Subject must be able to understand, read and sign the study specific informed consent forms after the nature of the study has been fully explained to her
3. Subject is indicated for myomectomy or polypectomy
4. Subject exhibits intrauterine polyps and/or submucous myomas which meet one of the following criteria. In cases of subjects with multiple intrauterine pathology, classification is based as follows:

   * All polyps
   * All Type 0, Type 1 or Type 2 myomas ≤ 6 cm in diameter
   * Polyps plus Type 0, Type 1 or Type 2 myomas ≤6 cm in diameter

Exclusion Criteria:

1. Subject is pregnant
2. Subject has an Intrauterine Device (IUD) at the time of the procedure. A subject may be enrolled in the study if the IUD is removed prior to the treatment procedure
3. Subject is taking an anticoagulant or antiplatelet medication other than low dose aspirin
4. Active pelvic inflammatory disease or pelvic/vaginal infection
5. Subject has a known or suspected coagulopathy or bleeding disorder
6. Subject has a history of disease which increases the risk for fluid overload (i.e. significant cardiac, hepatic, or renal dysfunction)
7. Subject has other co-morbid condition(s) that, in the opinion of the Investigator, could limit the subject's ability to participate in the study or impact the scientific integrity of the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Evantash, Principal Investigator — Hologic, Inc.
Locations (1):
- Hologic, Inc., Marlborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intrauterine Pathology, Myomectomy
Started | 290
Completed | 290
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 290 Subjects enrolled. Nine (9) subjects removed from analysis because they did not meet the inclusion criteria. Three (3) subjects removed from analysis because they met the exclusion criteria.
Arm/Group | Intrauterine Pathology, Myomectomy
Number analyzed (Participants) | 278
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 278
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 278

OUTCOME MEASURES:

1. Primary Outcome: Procedure Efficacy
Description: Mean percent of pathology removed, based on hysteroscopic assessment immediately following completion of the treatment procedure
Time Frame: 1 hour post treatment
Population: 559 pathologies, 187 Fibroids and 372 polyps, were removed from 278 patients.
Measure: Mean (95% Confidence Interval); unit: percent of pathology
Arm/Group | Intrauterine Pathology, Myomectomy
Number analyzed (Participants) | 278
percent of pathology | 95.4 [93.8 to 96.9]

2. Secondary Outcome: Percentage of Subjects That Achieve 100% Removal of Target Pathology
Description: Percentage of subjects that achieve 100% removal of target pathology, as determined by hysteroscopic exam following the treatment procedures.
Time Frame: 1 hour post treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intrauterine Pathology, Myomectomy
Number analyzed (Participants) | 278
percentage of participants | 74.6 [69.5 to 79.8]

ADVERSE EVENTS:
Arm/Group | Intrauterine Pathology, Myomectomy
Serious Adverse Events (participants affected / at risk) | 0/278
Other Adverse Events (participants affected / at risk) | 5/278
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrauterine Pathology, Myomectomy (N=278)
Cervical Trauma (Reproductive system and breast disorders) | 4 (4)
Pedal Edema Post-operative (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No